CLINICAL TRIAL: NCT00093171
Title: An Open-label Safety and Efficacy Study of Recombinant Human Factor IX (rFIX; BeneFIX®) in Previously Treated Patients (PTPs) With Hemophilia B (FIX:C ≤2%)
Brief Title: Study Evaluating rFIX; BeneFIX® in Hemophilia B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 3090A1-302
Record Dates: First submitted 2004-10-04; First posted 2004-10-07 (Estimated); Last update posted 2009-08-21 (Estimated); Status verified 2009-08

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B

INTERVENTIONS:
Drug: rFIX

SUMMARY:
The primary objective of this clinical research study is to assess the safety and efficacy of rFIX for a minimum of 6 months in previously treated patients (PTPs) with hemophilia B (FIX:C ≤2%) during standard-of-care treatment (on-demand, prophylaxis, and through major and minor surgical procedures).

ELIGIBILITY:
Inclusion Criteria:

* Hemophilia B (FIX:C less than 2%)
* Previous treatment of at least 150 exposure days using any FIX product
* 12 years of age and older

Exclusion Criteria:

* The patient has a currently detectable factor IX inhibitor or a history of inhibitors. (A family history of inhibitors will not exclude the patient)
* Known hypersensitivity to protein pharmaceuticals or agents related to the test article, e.g. hamster proteins
* Patient has a genetic coagulation disorder other than hemophilia B

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (7):
- United States (7):
  - Los Angeles, California
  - Aurora, Colorado
  - Detroit, Michigan
  - New Brunswick, New Jersey
  - Chapel Hill, North Carolina
  - Dayton, Ohio
  - Houston, Texas

REFERENCES:
- [Derived] Wojciechowski J, Gaitonde P, Hughes JH, Ravva P. Population Modeling of Factor IX Activity Following Administration of Fidanacogene Elaparvovec Gene Therapy in Participants with Hemophilia B. Clin Pharmacokinet. 2025 Oct;64(10):1531-1548. doi: 10.1007/s40262-025-01535-y. Epub 2025 Aug 1. PMID 40750723
- [Derived] Rendo P, Smith L, Lee HY, Shafer F. Nonacog alfa: an analysis of safety data from six prospective clinical studies in different patient populations with haemophilia B treated with different therapeutic modalities. Blood Coagul Fibrinolysis. 2015 Dec;26(8):912-8. doi: 10.1097/MBC.0000000000000359. PMID 26196195